CLINICAL TRIAL: NCT01794702
Title: Phase I/II Study of Decitabine (DAC) Followed by Clofarabine, Idarubicin, and Cytarabine (CIA) in Acute Leukemia
Brief Title: Decitabine Followed by Clofarabine, Idarubicin, and Cytarabine in Acute Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2012-1064; NCI-2013-00548 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-02-15; First posted 2013-02-20 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Leukemia
Keywords: Leukemia; Acute Leukemia; Acute myelogenous leukemia; AML; Acute lymphoblastic leukemia; ALL; Maximum Tolerated Dose; MTD; Response Rate; Decitabine; Dacogen; Idarubicin; Idamycin; Cytarabine; Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Decitabine; Idarubicin; Cytarabine; Clofarabine

STUDY DESIGN:
Intervention Model Description: Starting with Dose level 1, the participants were enrolled by cohort of 3. Once the DLT assessment is completed, another cohort of 3 patients will be enrolled. If at any time, we see more than 30% patients experiencing DLT, we will de-escalate to dose level (-1).
  Period 1: Dose level 1 Clofarabine 15mg/m^2 daily x 4 days (days 6-9)
  Period 2: Dose level-1 Clofarabine 15mg/m^2 daily x 3 days (days 6-8)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Clofarabine + Cytarabine + Decitabine + Idarubicin (Experimental): Phase I - Decitabine 20 mg/m2 by vein over approximately 1 hour daily for 5 days (days 1-5) Idarubicin 10 mg/m2 by vein over approximately 30 minutes daily for 3 days (days 6-8) Cytarabine 1 g/m2 by vein over approximately 2 hours daily for 5 days (days 6-10)
  Phase II - Clofarabine 15 mg/m2 by vein over approximately 1 hour daily (number of days selected based on Phase I portion).
  Decitabine 20 mg/m2 by vein over approximately 1 hour daily for 5 days (days 1-5) Idarubicin 10 mg/m2 by vein over approximately 30 minutes daily for 3 days (days 6-8) Cytarabine 1 g/m2 by vein over approximately 2 hours daily for 5 days (days 6-10)
  Interventions: Drug: Decitabine; Drug: Idarubicin; Drug: Cytarabine; Drug: Clofarabine

INTERVENTIONS:
Drug: Decitabine — Phase I and II - 20 mg/m2 by vein daily for 5 days (days 1-5)
  Other Names: Dacogen
Drug: Idarubicin — Phase I and II - 10 mg/m2 by vein daily for 3 days (days 6-8)
  Other Names: Idamycin
Drug: Cytarabine — Phase I and II - 1 g/m2 by vein daily for 5 days (days 6-10)
  Other Names: Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
Drug: Clofarabine — Phase I Starting Dose - 15 mg/m2 by vein daily for 4 days (days 6-9)
  Phase II Starting Dose - Maximum tolerated dose from Phase I (number of days selected based on Phase I portion).
  Other Names: Clofarex; Clolar

SUMMARY:
The goal of Phase I of this clinical research study is find the highest tolerable dose of clofarabine that can be given with decitabine, idarubicin, and cytarabine to patients with acute leukemia.

The goal of Phase II of this study is to learn if decitabine followed by the combination of clofarabine, idarubicin, and cytarabine can help to control acute leukemia. The safety of this drug combination will also be studied.

Decitabine and idarubicin are designed to damage the DNA (the genetic material of cells). This may cause cancer cells to die.

Clofarabine is designed to interfere with the growth and development of cancer cells.

Cytarabine is designed to insert itself into DNA and stop the DNA from repairing itself.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 3 groups of 6 participants will be enrolled in the Phase I portion of the study. Up to 74 participants will be enrolled in Phase II.

Phase I:

If you are enrolled in the Phase I portion, the number of days of clofarabine you receive will depend on when you joined this study. The first group of participants will receive clofarabine for 4 days. Each new group will receive clofarabine for the same number of days, if no intolerable side effects were seen. The number of days may be reduced to 3. The clofarabine dose per day is the same from group to group.

All participants will receive the same dose level of decitabine, idarubicin and cytarabine.

Phase II:

If you are enrolled in the Phase II portion, you will receive decitabine, idarubicin, and cytarabine. You will receive clofarabine for the highest number of days that was tolerated in the Phase I portion.

All participants will receive the same dose level of decitabine, idarubicin, cytarabine, and clofarabine.

Study Drug Administration:

Each study drug cycle is 33 days. The first cycle of study drugs is called Induction. If the doctor thinks it is needed, you will have up to 2 Induction cycles.

Phase I (Induction):

On Days 1-5 of each cycle, you will receive decitabine 1 time a day by vein over about 1 hour.

On Days 6-10 of each cycle:

* You will receive cytarabine 1 time a day by vein over about 2 hours.
* On Days 6-8 only, you will receive idarubicin 1 time a day by vein over about 30 minutes.
* You will receive clofarabine 1 time a day by vein over about 1 hour on Days 6-8 or 6-9, depending on when you join the study.

If the doctor thinks it is needed, your dose level will be reduced after Induction.

If the doctor thinks it is needed, you may receive fewer days of treatment in the Induction cycle(s).

Phase II (Induction):

On Days 1-5 of each cycle, you will receive decitabine 1 time a day by vein over about 1 hour.

On Days 6-10 of each cycle:

* You will receive cytarabine 1 time a day by vein over about 2 hours.
* On Days 6-8 only, you will receive idarubicin 1 time a day by vein over about 30 minutes.
* You will receive clofarabine 1 time a day by vein over about 1 hour on Days 6-8 or 6-9, depending on the highest number of days clofarabine was tolerated in the Phase I portion of the study.

If the doctor thinks it is needed, your dose level will be reduced after Induction.

If the doctor thinks it is needed, you may receive fewer days of treatment in the Induction cycle(s).

Phases I and II (Consolidation):

If the disease responds to the study drugs, you may receive up to 6 more study drug cycles. This is called Consolidation.

On Days 1-5 of each cycle:

°You will receive decitabine 1 time a day by vein over 1 hour.

On Days 6-8 of each cycle:

* You will receive cytarabine 1 time a day by vein over about 2 hours.
* You will receive clofarabine 1 time a day by vein over about 1 hour.
* On Days 6-7 only, you will receive idarubicin 1 time a day by vein over about 30 minutes.

If the doctor thinks it is needed, you may receive fewer days of treatment in the Consolidation cycles.

Study Visits:

Before the start of each cycle, you will have a physical exam, including measurement of your vital signs.

Every 3-7 days, blood (about 2 teaspoons) will be drawn for routine tests.

On Day 33 of every 2-3 cycles (+/- 7 days), if the doctor thinks it is needed, you will have a bone marrow aspirate to check the status of the disease. To collect a bone marrow aspirate, an area of the hip is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle.

Length of Treatment:

You may continue taking the study drugs for up to 8 cycles. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the long-term follow-up.

Long-term Follow-up:

Every 3 months for 1 year after your last study drug dose, the study staff will call you and ask how you are feeling, about any side effects you may be having, and about any other drugs you may be taking. These calls should last about 5 minutes each.

This is an investigational study. Decitabine is FDA approved and commercially available to treat myelodysplastic syndrome (MDS). Clofarabine is FDA approved and commercially available to treat ALL in children. Idarubicin and cytarabine are FDA approved and commercially available to treat AML. The study drug combination is investigational.

Up to 92 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an IRB-approved informed consent document.
2. Age >/= 18 years and <65 years.
3. Diagnosis of AML [other than acute promyelocytic leukemia] with refractory/relapsed disease (Patients must be primary refractory, in relapse 1, or in relapse 2). NOTE: Patients with AML arising from prior MDS or MPN would be eligible even if they have not received treatment for the AML. NOTE: Patients with relapsed/refractory ALL would also be eligible for the phase II part of the study. NOTE: Use of hydroxyurea and/or up to 4 doses of cytarabine, for emergent cytoreduction is allowed
4. ECOG performance status of </=2 at study entry.
5. Organ function as defined below (unless due to leukemia):Serum creatinine </= 3 mg/dL;Total bilirubin </= 2.5 mg/dL; ALT (SGPT) </= 3 x ULN or </= 5 x ULN if related to disease
6. Cardiac ejection fraction ≥ 40% (by either cardiac ECHO or MUGA scan)
7. Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential.

Exclusion Criteria:

1. Breast feeding women
2. Patients with uncontrolled active infections (viral, bacterial, and fungal are not eligible).
3. Patients with active secondary malignancy will not be eligible unless approved by the PI.
4. NOTE: Prior therapy with decitabine, clofarabine, idarubicin, or cytarabine is allowed, unless the prior therapy is identical to the schema/schedule proposed in this study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2013-02-20 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Jain, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 1/2013 to 01/2018
Pre-assignment Details: All participants in the phase I portion of the study received dose level 1 of the study medication. None of the participants experienced a DLT as defined in the protocol.
  Period 1: Dose level 1 - Clofarabine 15mg/m^2 daily x 4 days (days 6-9) Period 2: Dose level-1 - Clofarabine 15mg/m^2 daily x 3 days (days 6-8)
Groups:
- Period 1: Phase I Clofarabine + Cytarabine + Decitabine + Idarubicin
  Phase I - Decitabine 20 mg/m^2 by vein for approximately 1 hour daily for 5 days (days 1-5) Idarubicin 10 mg/m^2 by vein for approximately 30 minutes daily for 3 days (days 6-8) Cytarabine 1 g/m^2 by vein for approximately 2 hours daily for 5 days (days 6-10)
  Clofarabine: Phase I Starting Dose - 15 mg/m^2 by vein daily for 4 days (days 6-9)
- Period 2: Phase I Clofarabine + Cytarabine + Decitabine + Idarubicin
  Phase I - Decitabine 20 mg/m^2 by vein for approximately 1 hour daily for 5 days (days 1-5) Idarubicin 10 mg/m^2 by vein for approximately 30 minutes daily for 3 days (days 6-8) Cytarabine 1 g/m^2 by vein for approximately 2 hours daily for 5 days (days 6-10)
  Clofarabine: Phase I Dose level -1 - 15 mg/m^2 by vein daily for 3 days (days 6-9)
- Phase II Clofarabine + Cytarabine + Decitabine + Idarubicin: Phase II - Decitabine 20 mg/m^2 by vein for approximately 1 hour daily for 5 days (days 1-5) Idarubicin 10 mg/m^2 by vein for approximately 30 minutes daily for 3 days (days 6-8) Cytarabine 1 g/m^2 by vein for approximately 2 hours daily for 5 days (days 6-10)
  Phase II - Clofarabine 15 mg/m^2 by vein over approximately 1 hour for 4 days (days 6-9).
Period: Overall Study
Arm/Group | Period 1 | Period 2 | Phase II Clofarabine + Cytarabine + Decitabine + Idarubicin
Started | 18 | 0 | 47
Completed | 18 | 0 | 47
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants in the phase I portion of the study received dose level 1 of the study medication. None of the participants experienced a DLT as defined in the protocol.
  Period 1 Dose level 1 - Clofarabine 15mg/m^2 daily x 4 days (days 6-9) Period 2 Dose level-1 - Clofarabine 15mg/m^2 daily x 3 days (days 6-8)
Groups:
- Period 2: Phase I Clofarabine + Cytarabine + Decitabine + Idarubicin
  Phase I - Decitabine 20 mg/m^2 by vein for approximately 1 hour daily for 5 days (days 1-5) Idarubicin 10 mg/m^2 by vein for approximately 30 minutes daily for 3 days (days 6-8) Cytarabine 1 g/m^2 by vein for approximately 2 hours daily for 5 days (days 6-10)
  Clofarabine: Phase I Dose -1 - 15 mg/m^2 by vein daily for 3 days (days 6-9)
- Phase II Clofarabine + Cytarabine + Decitabine + Idarubicin: Phase II - Decitabine 20 mg/m^2 by vein for approximately 1 hour daily for 5 days (days 1-5) Idarubicin 10 mg/m^2 by vein for approximately 30 minutes daily for 3 days (days 6-8) Cytarabine 1 g/m^2 by vein for approximately 2 hours daily for 5 days (days 6-10)
  Phase II - Clofarabine 15 mg/m2 by vein over approximately 1 hour for 4 days (days 6-9).
- Total: Total of all reporting groups
Arm/Group | Period 1 | Period 2 | Phase II Clofarabine + Cytarabine + Decitabine + Idarubicin | Total
Number analyzed (Participants) | 18 | 0 | 47 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 0 | 47 | 65
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 15 | 18
  Male | 15 | 0 | 32 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 8 | 9
  White | 14 | 0 | 33 | 47
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 18 |  | 47 | 65

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Clofarabine
Description: Maximum tolerated dose (MTD) defined as the highest dose schedule in which 6 patients were treated with at most 1 experiencing a dose-limiting toxicity (DLT). Clofarabine 15 mg/m2 IV over approximately 1 hour daily (number of days selected based on Phase I portion).
Time Frame: After second, 33 day cycle
Population: All participants in the phase I portion of the study received dose level 1 of the study medication. None of the participants experienced a DLT as defined in the protocol.
  Period 1: Dose level 1 - Clofarabine 15mg/m^2 daily x 4 days (days 6-9) Period 2: Dose level-1 - Clofarabine 15mg/m^2 daily x 3 days (days 6-8)
Measure: Number; unit: mg/m^2 x 4 days (6-9)
Groups:
- Period 1; Period 2: Clofarabine + Cytarabine + Decitabine + Idarubicin
  Phase I - Decitabine 20 mg/m^2 by vein over approximately 1 hour daily for 5 days (days 1-5) Idarubicin 10 mg/m^2 by vein over approximately 30 minutes daily for 3 days (days 6-8) Cytarabine 1 g/m^2 by vein over approximately 2 hours daily for 5 days (days 6-10)
  Clofarabine 15 mg/m^2 by vein over approximately 1 hour daily
Arm/Group | Period 1 | Period 2
Number analyzed (Participants) | 18 | 0
mg/m^2 x 4 days (6-9) | 15 |

2. Primary Outcome: Number of Participants With a Response
Description: Primary endpoint is overall response defined as the best response either complete response, complete remission without platelet recovery, or complete remission without incomplete blood count recovery within 56 days.
Time Frame: 56 days
Population: One of the 47 participants on the Phase II portion of this study who received study medication was not evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II Clofarabine + Cytarabine + Decitabine + Idarubicin
Number analyzed (Participants) | 46
Participants | 20

3. Secondary Outcome: To Determine the Disease-free Survival (DFS).
Description: Time from date of treatment start until the date of first objective documentation of return of disease.
Time Frame: Up to 2 years after participants off study date
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | Phase II Clofarabine + Cytarabine + Decitabine + Idarubicin
Number analyzed (Participants) | 46
months | 17.9 [1 to 33]

4. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 2 years after participants off study date
Population: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | Phase II Clofarabine + Cytarabine + Decitabine + Idarubicin
Number analyzed (Participants) | 46
Months | 7.7 [1 to 40]

ADVERSE EVENTS:
Time Frame: 3 years
Description: All participants in the phase I portion of the study received dose level 1 of the study medication. None of the participants experienced a DLT as defined in the protocol.
  Period 1 Dose level 1 - Clofarabine 15mg/m^2 daily x 4 days (days 6-9) Period 2 Dose level-1 - Clofarabine 15mg/m^2 daily x 3 days (days 6-8)
Arm/Group | Period 1 | Period 2 | Phase II Clofarabine + Cytarabine + Decitabine + Idarubicin
All-Cause Mortality (participants affected / at risk) | 1/18 | 0/0 | 5/46
Serious Adverse Events (participants affected / at risk) | 18/18 | 0/0 | 33/46
Other Adverse Events (participants affected / at risk) | 17/18 | 0/0 | 27/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1 (N=18) | Period 2 (N=0) | Phase II Clofarabine + Cytarabine + Decitabine + Idarubicin (N=46)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | NA | 0 (0)
Death (General disorders) | 1 (1) | NA | 0 (0)
Elevated Transaminases (Metabolism and nutrition disorders) | 3 (5) | NA | 0 (0)
Gastric Hemorrhage (Blood and lymphatic system disorders) | 1 (1) | NA | 0 (0)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 2 (2) | NA | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | NA | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | NA | 1 (1)
Left Ventricular Failure (Cardiac disorders) | 1 (1) | NA | 0 (0)
Mucositis (Gastrointestinal disorders) | 2 (2) | NA | 0 (0)
Neutropenic Fever (Infections and infestations) | 13 (24) | NA | 24 (38)
Pain (General disorders) | 3 (4) | NA | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | 0 (0)
Seizures (Nervous system disorders) | 1 (1) | NA | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | NA | 1 (1)
Septic Shock (Infections and infestations) | 2 (2) | NA | 1 (1)
Abcess (Skin and subcutaneous tissue disorders) | 0 (0) | NA | 1 (1)
Bronchopulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | NA | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | NA | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | NA | 1 (1)
Headache (General disorders) | 0 (0) | NA | 1 (1)
Infection (Infections and infestations) | 0 (0) | NA | 1 (1)
Intracranial Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | NA | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | NA | 1 (1)
Neutropenia (Infections and infestations) | 0 (0) | NA | 1 (1)
Typhlitis (Gastrointestinal disorders) | 0 (0) | NA | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1 (N=18) | Period 2 (N=0) | Phase II Clofarabine + Cytarabine + Decitabine + Idarubicin (N=46)
Infection (Infections and infestations) | 1 (1) | NA | 5 (5)
Mucositis (Gastrointestinal disorders) | 2 (2) | NA | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (5) | NA | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 13 (13) | NA | 15 (17)
Elevated Transaminases (Metabolism and nutrition disorders) | 10 (10) | NA | 13 (14)
Nausea (Gastrointestinal disorders) | 3 (3) | NA | 0 (0)
Pain (General disorders) | 2 (2) | NA | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | NA | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | NA | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | NA | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT01794702/Prot_SAP_000.pdf